CLINICAL TRIAL: NCT03889808
Title: Seroprevalence of Anti-bodies Against Clostridium Difficile Toxins and Prevalence of Asymptomatic Carriage of Clostridium Difficile in IBD Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Claudia Arajol Gonzalez, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: JGC-INM-2014-01
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Clostridium Difficile; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Non immunosuppressed patients: without treatment or treated with Salicylates and that have not received immunosuppressive therapy, steroids, or biologics in the last 6 months.
  Interventions: Diagnostic Test: Determination of serum anti-toxin Abs for C. difficile
- Patients with immunosuppressive therapy: Azathioprine, 6-Mercaptopurine, Methotrexate in standard dosage at least the past 6 months and that have not received steroids or biologics in the last 6 months.
  Interventions: Diagnostic Test: Determination of serum anti-toxin Abs for C. difficile
- Patients with biologic agents: in standard dosage at least the past 6 months and that have not received steroids in the previous 6 months.
  Interventions: Diagnostic Test: Determination of serum anti-toxin Abs for C. difficile
- Patients with steroid treatment: Must have received daily steroid treatment ≥ 20 mg for ≥ 2 weeks.
  Interventions: Diagnostic Test: Determination of serum anti-toxin Abs for C. difficile
- Healthy subjects: A healthy subject is defined as not having and immunosuppressive underlying condition, not receiving immunosuppressive therapy, has not received antibiotic treatment in the last 6 months, has no past C. difficile infections and has not been in contact with the health care system or hospitalized in the previous 6 months.
  Interventions: Diagnostic Test: Determination of serum anti-toxin Abs for C. difficile

INTERVENTIONS:
Diagnostic Test: Determination of serum anti-toxin Abs for C. difficile
  Other Names: Stool culture for C. difficile

SUMMARY:
The objective of this study to evaluate the seroprevalence of anti-bodies against C. difficile toxins A and B and the asymptomatic carriage of C. difficile in IBD patients according to the need and type of immunosuppressive therapy. The ultimate goal is to identify, among IBD patients, those with the highest risk of CDI.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosed of IBD, either Crohn's disease or ulcerative colitis
* Age: >18 and <65 years
* Time since diagnoses of IBD ≥ 6 months
* Present with the criteria included in any of the 4 specified groups in the study population

Exclusion Criteria:

* History of documented CDI
* Active CDI at the moment of study inclusion
* Any of the following immunosuppressive conditions: HIV infection, Liver cirrhosis, CKD stage IV, Receiving chemotherapy, Transplant (solid organ or hematological), Concomitant neoplasia, Hypogammaglobinemia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study would include 400 patients with IBD (Crohn's disease and ulcerative colitis).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Clostridium difficile anti-toxin Abs in patients with IBD | 0 days
  Determination of serum anti-toxin Abs for C. difficile with ELISA (enzyme-linked immunosorbent assay). The concentration of C. difficile anti-toxin Abs will be categorized as: < 25 percentile: Low, >26 < 75 percentiles: Intermediate, >76 <90 percentiles: High, >91 percentile: Very high.
Prevalence of asymptomatic carrier of Clostridium difficile in patients with IBD | 0 days
  Stool testing for C. difficile as part of a multiple step algorithm: GDH (glutamate dehydrogenase), toxin EIA (enzyme immunoassay) test and C. difficile culture.
Study the relationship between the different maintenance therapies for IBD and C. difficile anti-toxin Abs and asymptomatic carriers. | 0 days

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Guardiola, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided